CLINICAL TRIAL: NCT00063297
Title: Safety and Efficacy of Study Drug Versus Placebo for Negative Symptoms of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004342
Record Dates: First submitted 2003-06-25; First posted 2003-06-26 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2003-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia with negative symptoms
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: R209130

SUMMARY:
This study is to determine the efficacy (how well the drug works), safety, and side effects of the study medication compared to placebo in the treatment of the negative symptoms of schizophrenia in adults.

ELIGIBILITY:
Inclusion:

* Adults aged 18-60
* Current diagnosis of schizophrenia
* Significant negative symptoms with few positive symptoms (e.g. hallucinations, delusions) and no evidence of major depression.
* Female subjects of childbearing potential must test negative for pregnancy at the time of enrollment.
* Subjects must be able to provide consent
* Must be healthy based on medical exam, laboratory tests and electrocardiogram

Exclusion:

* Female subjects who are either pregnant or nursing.
* Acute or unstable medical conditions
* Diseases of the central nervous system
* Subjects who are judged clinically to be at serious risk for suicide or violence
* Subjects with delusional disorder, psychotic disorder NOS, schizophreniform, schizoaffective disorder, bipolar disorder, attention deficit/hyperactivity disorder, major depressive disorder,alcohol or drug dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180
Dates: Start 2003-05; Study Completion 2003-10

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - IPR, Cerritos, California
  - Synergy Clinical Research, Chula Vista, California
  - Optimum Health Services, La Mesa, California
  - Sierra Vista Hospital, Sacramento, California
  - Clinical Innovations, Santa Ana, California
  - Research Strategies, Torrance, California
  - University of Colorado, Denver, Colorado
  - Psychiatric Institute of Washington, Washington D.C., District of Columbia
  - Berma Research Group, Hialeah, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Med Psych Specialists, LLC, Atlanta, Georgia
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - Midwest Center for Neurobehavioral Medicine, Oakbrook Terrace, Illinois
  - Shreveport, Louisiana
  - University of Mississippi Medical Center-Dept. of Psychiatry, Jackson, Mississippi
  - CNS Research Institute, Clementon, New Jersey
  - Neurobehavioral Research, Lawrence, New York
  - Global Research & Consulting, Olean, New York
  - Bayley Seton Campus-Psychiatric Research Division, Staten Island, New York
  - Behavioral Medical Research of Staten Island, P.C., Staten Island, New York
  - NorthCoast Clinical Trials, Beachwood, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Community Clinical Research, Austin, Texas
  - MedLabs Research of Houston, Houston, Texas
  - University Hills Clinical Research, Irving, Texas
  - Milwaukee VA Medical Center, Milwaukee, Wisconsin